CLINICAL TRIAL: NCT06659016
Title: EFFICACIA DI UN INTEGRATORE A BASE DI D-MANNOSIO, PROPOLI, QUERCETINA, COLLAGENE E BACILLUS COAGULANS NEL RIDURRE L'INCIDENZA E MIGLIORARE LA QUALITA' DI VITA IN DONNE CON CISTITE RICORRENTE
Brief Title: Efficacy of Collagen, Propolis Plus Quercetin (Proqutin®), Bacillus Coagulans, Hyaluronic Acid and Chondroitin Sulphate and D-Mannose to Avoid Symptoms and Prevents Recurrence in Women With Recurrent Urinary Tract Infections
Acronym: IMProBaCist-Q
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: pharmaSuisse (Unknown)
Responsible Party: Principal Investigator, Gaetano Riemma, Principal investigator, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10/2024/SCCAL
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Urinary Tract Infection (Diagnosis)
MeSH Terms: conditions — Urinary Tract Infections; Disease | interventions — Fosfomycin; alloxantin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are blind to treatment arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator)
  Interventions: Drug: Fosfomycin 3 g
- Group B (Experimental): Dietary supplement of D-mannose, collagen, hyaluronic acid, chondroitin sulphate, propolis plus quercetin (Proqutin ®) and Bacillus Coagulans (Uroxin 4G, Pharmasuisse laboratories, Milan, Italy) administered twice daily for seven days in the first month, then once daily for 14 days a month for two months, repeated every three months for a total treatment duration of 12 months.
  Interventions: Dietary Supplement: Uroxin 4G
- Group C (Experimental): Combination of treatment A and B
  Interventions: Drug: Combination of dietary supplement and fosfomycin

INTERVENTIONS:
Drug: Fosfomycin 3 g — Fosfomycin trometamol 3 g administered orally in a single dose every ten days for three months, repeated every three months for a total treatment duration of 12 months.
  Arms: Group A
Dietary Supplement: Uroxin 4G — Dietary supplement of D-mannose, collagen, hyaluronic acid, chondroitin sulphate, propolis plus quercetin (Proqutin ®) and Bacillus Coagulans (Uroxin 4G, Pharmasuisse laboratories, Milan, Italy) administered twice daily for seven days in the first month, then once daily for 14 days a month for two months, repeated every three months for a total treatment duration of 12 months.
  Arms: Group B
Drug: Combination of dietary supplement and fosfomycin — Fosfomycin trometamol 3 g administered orally in a single dose every ten days for three months, repeated every three months for a total treatment duration of 12 months, combined with an oral formulation of D-mannose, collagen, hyaluronic acid, chondroitin sulphate, propolis plus quercetin (Proqutin ®) and Bacillus Coagulans (Uroxin 4G, Pharmasuisse laboratories, Milan, Italy) administered twice daily for seven days in the first month, then once daily for 14 days a month for two months, repeated every three months for a total treatment duration of 12 months.
  Arms: Group C

SUMMARY:
The aim of this study is to evaluate whether a dietary supplement based on D-mannose, collagen, hyaluronic acid, chondroitin sulphate, enhanced by the properties of quercetin plus propolis (Proqutin ®) and Bacillus Coagulans, eventually associated with antimicrobial prophylaxis, could be effective in preventing recurrent UTIs and improving related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* a history of rUTIs (defined by EAU guidelines as a frequency of at least three UTIs per year, or two UTIs in the past six months in the last 12 months, confirmed by positive urine cultures
* not undergone any previous treatment for their condition.

Exclusion Criteria:

* age under or over limit
* concurrent antimicrobial treatment
* any ongoing treatment that could influence study outcomes,
* congenital or post-surgical urinary tract anomalies
* immunodeficiency or HIV infection
* ongoing pregnancy.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Number of urinary tract infections per month | 6 and 12 months

SECONDARY OUTCOMES:
ICIQ-FLUTS scores | 6 and 12 months
Number of women matching recurrent urinary tract infection criteria | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania Luigi Vanvitelli, Napoli, Italy

REFERENCES:
- [Derived] Riemma G, Vinci D, La Verde M, Caniglia FM, Scalzone G, Torella M. Adding collagen, propolis plus quercetin, bacillus coagulans, hyaluronic acid and chondroitin sulphate to D-mannose avoids symptoms and prevents recurrence in women with recurrent urinary tract infections: a single-blind randomized controlled trial. Expert Rev Anti Infect Ther. 2025 Jul;23(7):523-530. doi: 10.1080/14787210.2025.2487162. Epub 2025 Apr 3. PMID 40162673